CLINICAL TRIAL: NCT00644579
Title: bLAC - A Phase II Double-Blind, Placebo Controlled, Clinical Proof of Concept Trial of the Efficacy of 8 Weeks Treatment of Cutaneous Warts With bLAC in Immune Suppressed, Kidney Transplanted Patients
Brief Title: bLAC - Treatment of Cutaneous Warts in Immune Suppressed, Kidney Transplanted Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NatImmune A/S (Industry)
Responsible Party: NatImmune A/S, NatImmune
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-1205; EudraCT number: 2007-006738-33
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Cutaneous Warts
Keywords: wart; cutaneous; transplant; Cutaneous warts in immune suppressed, kidney transplant patients
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): bLAC high dose
  Interventions: Drug: bLAC
- 2 (Active Comparator): bLAC low dose
  Interventions: Drug: bLAC
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bLAC — bLAC high and low dose and placebo
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
As many as 85 % of renal transplant patients may suffer from viral warts with a high degree of treatment resistance. Promising results of hLAC (human lactalbumin complex with lipid) point to a beneficial effect without noticeable side effects of bLAC (bovine lactalbumin complex with lipid). The aim of first clinical trial with bLAC is to show proof of concept in treatment of cutaneous wart lesions on hands and/or feet after local administration of bLAC in two dose groups to immune suppressed, kidney transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous warts on ingers and/or palms and/or toes and/or soles of feet
* Common warts and mosaic warts, diagnosed by an experienced dermatologist
* Solitary wart lesions or 2 or more lesions per patient
* Lesions present for more than 6 months
* Men or women, aged 18 or above
* History of kidney transplantation and immune suppressive therapy after transplant
* Concomitant immune suppressive therapy stable for 6 months prior to randomization
* Agreement from patient to allow photographs to be taken and used as part of trial data documentation (2 centres)
* Women of childbearing potential must have negative pregnancy test at screening and must use adequate contraception
* Ability to comply with requirements of trial
* Written informed consent

Exclusion Criteria:

* Verruca plana lesions
* Suspected allergy to milk verified by serum analysis of IgE towards cow milk
* Breastfeeding
* Any local medication for any purpose other than wart treatment in target area during 4 weeks prior to randomization and during treatment period
* Concomitant treatment with other wart therapies two weeks prior to randomization and during trial period
* Intolerance towards bovine alpha-lactalbumin, oleic acid or any excipient in the formulation
* Known HIV infection or any current uncontrolled infection
* Any chronic or acute skin condition susceptible of interfering with evaluation of drug effect in this trial
* Participation in any investigational trial or use of any investigational drug within 30 days prior to inclusion in this trial
* Any health problems which according to Investigator's clinical judgment will make the patient unsuitable for inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in the area of wart lesions located on fingers and/or palms and/or toes and/or soles of the feet, measured by an objective method by drawing of individual lesions | Prospective

SECONDARY OUTCOMES:
Clearance of index wart lesions. Time to clearance of warts. Recurrence rate of previously cleared wart lesions. Occurrence of new warts.overall changes of index warts lesions. Safety and tolerability. | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Claus Zachariae, MD, Principal Investigator — Gentofte Amtssygehus
Locations (5):
- Denmark (5):
  - Dermatology Clinic, Vesterbro, Aalborg
  - Marselisborg University Hospital, Aarhus C
  - Bispebjerg University Hospital, Copenhagen NV
  - Gentoftte Amtssygehus, Hellerup
  - Odense University Hospital, Odense